CLINICAL TRIAL: NCT06229093
Title: Multimodal Musical Stimulation for Healthy Neurocognitive Aging
Acronym: Multimodal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Psyche Loui, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NortheasternMINDLabMultimodal
Record Dates: First submitted 2021-12-08; First posted 2024-01-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Aging
Keywords: Music
MeSH Terms: interventions — Electroencephalography Phase Synchronization

STUDY DESIGN:
Who Masked: Participant
Masking Description: The assignment of older adults to OA and OAg will be randomized. The within-subjects factor of stimulation modality includes 2 levels, to be administered in counterbalanced order: Visual (V, i.e., lights-only) and Audiovisual (AV, i.e., music-plus-lights). Each subject will be aware that they are receiving V and AV stimulation, and thus infer that we are comparing these two forms of stimulation and therefore assessing the effects of music. However, and important to the design of this study, all subjects will be blinded with respect to their group assignment; i.e., they will not know, until post-study debriefing, about the other arms of the study, and that the gamma-band stimulation is an active ingredient of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Adults (OA) (Sham Comparator): The assignment of older adults to OA and OAg will be randomized. The within-subjects factor of stimulation modality includes 2 levels, to be administered in counterbalanced order: Visual (V, i.e., lights-only) and Audiovisual (AV, i.e., music-plus-lights). Each subject will be aware that they are receiving V and AV stimulation, and thus infer that we are comparing these two forms of stimulation and therefore assessing the effects of music. However, and important to the design of this study, all subjects will be blinded with respect to their group assignment; i.e., they will not know, until post-study debriefing, about the other arms of the study, and that the gamma-band stimulation is an active ingredient of the intervention.
  Interventions: Device: Synchrony
- Older Adults Gamma (OAg) (Experimental): The assignment of older adults to OA and OAg will be randomized. The within-subjects factor of stimulation modality includes 2 levels, to be administered in counterbalanced order: Visual (V, i.e., lights-only) and Audiovisual (AV, i.e., music-plus-lights). Each subject will be aware that they are receiving V and AV stimulation, and thus infer that we are comparing these two forms of stimulation and therefore assessing the effects of music. However, and important to the design of this study, all subjects will be blinded with respect to their group assignment; i.e., they will not know, until post-study debriefing, about the other arms of the study, and that the gamma-band stimulation is an active ingredient of the intervention.
  Interventions: Device: Gamma

INTERVENTIONS:
Device: Gamma — For the OAg group, the visual component of multimodal stimulation will have the same properties as for the other group, except it will also be additionally amplitude-modulated in the gamma-band (30-60 Hz) range, resulting in a detectable flicker over-and-above the beat-level modulation.
  Arms: Older Adults Gamma (OAg)
Device: Synchrony — For the OA group, the lights will be tuned to delta-band frequencies (1-4 Hz) in the music, which corresponds to the beat-level frequency in most music. Thus, the lights automatically adapt to the rhythm of the music, pulsing on the beat and changing color on strong beats.
  Arms: Older Adults (OA)

SUMMARY:
This is a Stage I randomized, sham-controlled trial on the effects of multimodal musical stimulation on working memory in aging. Neurologically healthy older and younger adults will be tested on working memory and electroencephalography in the first randomized controlled trial of music as a form of brain stimulation, with multimodal musical stimulation and control stimulation conditions. Results will test the causal role of oscillatory mechanisms of the brain on cognition, and will lay the groundwork to the first musical, neurophysiologically targeted, brain-stimulation device for reversing cognitive decline in aging.

DETAILED DESCRIPTION:
Music contains amplitude and frequency modulations, rapid changes in acoustic signals that convey meaningful information to the listener. The human brain's ability to receive and interpret meaning from these signals is implemented by networks of neural oscillations: firing patterns of groups of neurons that track the music with rhythmic activity. Neural oscillations in different frequency bands subserve attention and memory, as well as perception and comprehension; they develop over the lifespan and are reduced in aging, especially in dementia. Being able to understand and causally control neural oscillations will have crucial implications for healthy neurocognitive aging. Since music naturally stimulates the brain with its rhythmic content over time, music may be used as a sustainable, naturalistic form of brain stimulation to induce oscillatory in neuronal populations. Furthermore, by inserting gamma-band energy as sensory stimulation during music listening, gamma-band activity may be increased in the brain in a way that is frequency-tuned to the brain's intrinsic network dynamics, thus replacing the decreased neural oscillations that are reduced in aging, and improving memory and cognition in older adults. The hypothesis is that gamma-band modulations inserted in lights, when coupled with music listening, can improve memory in older adults by frequency-tuning to intrinsic individual brain network dynamics. Results will test the causal role of oscillatory mechanisms of the brain on cognition. If successful, this trial will lay the groundwork to the first musical, neurophysiologically targeted, brain-stimulation device for reversing cognitive decline in aging.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected-to-normal vision
* no more than mild hearing loss
* no recent history of neurological or psychiatric disorders, including mood disorders or use of medications that may affect cognition or responsiveness to music.

Exclusion Criteria:

* moderate or severe hearing loss (40+ dB)
* visual impairment (including color blindness) that cannot be corrected with glasses or contacts
* recently changed dosage of cholinesterase inhibitors or psychotropic medication
* recent history of psychotic or schizophrenic episodes
* major neurologic diagnosis or other condition that might impair cognition or confound assessments (dementia, ADRD; Parkinson's disease, stroke, brain injury, epilepsy, or recent cardiovascular or neurovascular event)
* recent history of serious physical trauma or diagnosis of serious chronic health condition requiring medical treatment and monitoring .

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
EEG | 8 weeks
  Delta, theta, and gamma frequencies

SECONDARY OUTCOMES:
Working Memory | 8 weeks
  delayed-matched-to-sample task

CONTACTS AND LOCATIONS:
Overall Officials: Psyche Loui, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No